CLINICAL TRIAL: NCT04366713
Title: An Open-Label Phase 2 Study to Characterize Colon Pathology in Patients With HER2 Amplified Breast Cancer Treated With Neratinib
Brief Title: A Study to Characterize Colon Pathology in Patients With HER2 Amplified Breast Cancer Treated With Neratinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PUMA-NER-6203; 2019-001896-35 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-04-29 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: HER2 Amplified Breast Cancer
Keywords: HER2-Positive; Breast Cancer; Colon Pathology; Colonoscopy
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Capecitabine; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neratinib (Experimental): Neratinib with loperamide prophylaxis, and capecitabine for participants treated for metastatic breast cancer
  Interventions: Drug: Neratinib; Drug: Capecitabine; Drug: Loperamide

INTERVENTIONS:
Drug: Neratinib — Administered orally once daily as a single daily dose of 240 mg
  Other Names: Nerlynx
Drug: Capecitabine — Administered orally twice daily at 750 mg/m^2 for 14 days of each 21 day treatment cycle
Drug: Loperamide — Administered orally for prophylaxis for 28 days and then as needed

SUMMARY:
This study will investigate colon pathology in patients with HER2-positive breast cancer treated with neratinib. Colonoscopy will be performed after eligibility has been confirmed, prior to administration of the first dose of neratinib, and after 28 days of neratinib treatment.

DETAILED DESCRIPTION:
This is an open-label, phase 2 study that will investigate colon pathology in patients with HER2-positive breast cancer treated with neratinib as monotherapy.

All patients will receive neratinib for the first 28 days as a single daily dose of 240 mg.

Colonoscopy will be performed after eligibility has been confirmed, but prior to administration of the first dose of neratinib and at Day 30 (± 3 days) the conclusion of Cycle 1 (28 days).

Following the second study colonoscopy procedure:

* For patients being treated for stage 1 to 3c breast cancer in the extended adjuvant setting, neratinib will continue to be administered at a single daily dose of 240 mg until completion of one year of therapy from start of treatment, or until disease recurrence (as determined by the Investigator), death, unacceptable toxicity, or other specified withdrawal criterion.
* For patients being treated for metastatic breast cancer (mBC), capecitabine will be introduced after the second study colonoscopy procedure at a dose of 750mg/m2 twice daily for 14 days of each 21 day treatment cycle, with neratinib administered continuously throughout at 240 mg daily, until disease progression, death, unacceptable toxicity, or other specified withdrawal criterion.

All patients will receive loperamide diarrhea prophylaxis daily for one 28-day cycle and then as needed.

ELIGIBILITY:
INCLUSION CRITERIA

1. Aged ≥18 years.
2. Histologically confirmed stage 1 through stage 4 primary adenocarcinoma of the breast.
3. Documented HER2 overexpression or gene-amplified tumor by a validated approved method.
4. Participants with confirmed stage 1 to stage 3c breast cancer receiving extended adjuvant treatment with neratinib monotherapy must have completed a course of prior adjuvant trastuzumab or experienced side effects that resulted in early discontinuation of trastuzumab that have since resolved.
5. Participants with mBC must have had at least 2 prior HER2-directed regimens.
6. Left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
7. Eastern Cooperative Oncology Group (ECOG) status of 0 to 1.
8. Negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause. [Women are considered postmenopausal if they are ≥12 months without menses, in the absence of endocrine or anti-endocrine therapies.]
9. Women of childbearing potential must agree and commit to the use of a highly effective non-hormonal method of contraception, i.e., intrauterine device, bilateral tubal ligation, vasectomized partner, or abstinence (only when it is the preferred lifestyle of the participant), from the time of informed consent until 28 days after the last dose of the investigational products. Men (male participant) with a female partner of childbearing potential must agree and commit to use condom and the female partner must agree and commit to use a highly effective method of contraception (i.e., any of the above methods, or for females, hormonal contraception associated with inhibition of ovulation) while on treatment and for 3 months after last dose of investigational products.
10. Recovery (i.e., to Grade 1 or baseline) from all clinically significant adverse events related to prior therapies (excluding alopecia, neuropathy, and nail changes).
11. No major bleeding diathesis or use of anticoagulants that would pose a high risk for endoscopic procedure.
12. Provide written, informed consent to participate in the study and follow the study procedures.

EXCLUSION CRITERIA:

1. Participants with confirmed stage 1 to stage 3c currently receiving chemotherapy, radiation therapy, immunotherapy, or biotherapy for breast cancer.
2. Participants with mBC who have received prior capecitabine or HER2 directed tyrosine kinase inhibitor (TKI) therapy.
3. Currently using drugs that have been implicated as causing microscopic colitis/watery diarrhea, such as acarbose, aspirin, proton pump inhibitors, nonsteroidal anti-inflammatory drugs (NSAIDs), histamine H2 receptor antagonists, selective serotonin reuptake inhibitors, and ticlopidine (Pardi, 2017).
4. Major surgery within <28 days of starting treatment or received chemotherapy, investigational agents, or other cancer therapy, except hormonal therapy (e.g., tamoxifen, aromatase inhibitors), <14 days prior to the initiation of investigational products.
5. Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2; including individuals who currently use digitalis, beta-blockers, or calcium channel blockers specifically for congestive heart failure), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia.
6. Corrected QT Interval (QTc) interval >0.450 seconds (males) or >0.470 (females), or known history of QTc prolongation or Torsade de Pointes (TdP).
7. Diagnosis of inflammatory bowel disease
8. Screening laboratory assessments outside the following limits:

   Laboratory Parameters Required Limit for Exclusion Absolute neutrophil count (ANC) <1,000/µl (<1.0 x 109/L) Platelet count <50,000/µl (<100 x 109/L) Hemoglobin <8 g/dL (transfusions allowed) Transfusions must be at least 14 days prior to initiation of treatment Total bilirubin >1.5 x institutional upper limit of normal (ULN) (in case of known Gilbert's syndrome, <2 x ULN is allowed) Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x institutional ULN (>5 x ULN if liver metastases are present) Creatinine Creatinine clearance <30 mL/min (as calculated by Cockcroft-Gault formula A or Modification of Diet in Renal Disease formula B) International Normalized Ratio (INR) >1.5 a Cockcroft and Gault, 1976 b Levey et al, 1999
9. Active, unresolved infections.
10. Participants with a second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Participants with other non-mammary malignancies must have been disease free for at least 5 years.
11. Currently pregnant or breast-feeding.
12. Significant chronic gastrointestinal disorder with diarrhea as a major symptom (eg, Crohn's disease, malabsorption, or Grade ≥2 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE v.4.0] diarrhea of any etiology at baseline).
13. Clinically active infection with hepatitis B or hepatitis C virus.
14. Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that could, in the Investigator's judgment, make the person inappropriate for this study.
15. Known hypersensitivity to any component of the investigational products; known allergies to any of the medications or components of medications used in the trial.
16. Unable or unwilling to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Puma Biotechnology, Inc.
Locations (1):
- Hospital CUF Descobertas, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with stage 1 to 3c disease receiving extended adjuvant therapy are anticipated to participate in the study for approximately 1 year: 1 month for screening and 12 months of treatment, and 1 month of safety follow up.
  Patients with mBC are anticipated to participate in the study for an average of 12 month: 1 month of screening, 9.5 months for treatment, and 1 month of safety follow up.
Pre-assignment Details: Screening activities are to be conducted within 28 days prior to Cycle 1/Day 1, except for serum or urine pregnancy test for women of child-bearing potential, which should be performed, both, at screening and repeated within 72 hours prior to Cycle 1/Day 1.
  Documentation of locally assessed ERBB2-amplified status by fluorescence in situ hybridization (FISH) (>2.2) or ERBB2 overexpression by immunohistochemistry (IHC) (3+) by a validated approved method (Wolff et al, 2013) must be confirmed.
Groups:
- Breast Cancer Participants Treated With Neratinib: Participants with stage 1 to 3c disease receiving extended adjuvant therapy are anticipated to participate in the study for approximately 1 year: 1 month for screening and 12 months of treatment, and 1 month of safety follow up.
  Patients with mBC are anticipated to participate in the study for an average of 12 month: 1 month of screening, 9.5 months for treatment, and 1 month of safety follow up.
Period: Overall Study
Arm/Group | Breast Cancer Participants Treated With Neratinib
Started | 6
Treated | 5
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Safety population (treated patients)
Groups:
- Neratinib: Overall Neratinib all arms
Arm/Group | Neratinib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Colon Pathology
Description: The primary endpoint is to describe the changes in colon pathology between the baseline colonoscopy and the second colonoscopy.
Time Frame: From baseline to second colonoscopy, which is 88 days after start of neratinib treatment.
Population: Subjects who had a baseline colonoscopy and a second colonoscopy with findings to report.
Measure: Number; unit: participants
Groups:
- Neratinib Patients With 2 Colonoscopies: Subjects who had a baseline colonoscopy and a second colonoscopy with findings to report.
Arm/Group | Neratinib Patients With 2 Colonoscopies
Number analyzed (Participants) | 4
participants
  No Significant Findings | 2
  Mild Changes | 2

2. Secondary Outcome: Incidence and Severity of Diarrhea
Description: Incidence and severity of treatment emergent (TEAE) diarrhea will be summarized according to the NCI-CTCAE version 4.0 in the first cycle of neratinib treatment, which is from the time of the first colonoscopy to the second colonoscopy, or 28 days for subjects with only one colonoscopy. Incidence is defined as the number of patients experiencing diarrhea divided by the number of patients at risk.
Time Frame: From baseline to second colonoscopy, which is 88 days after start of neratinib treatment.
Population: All treated patients
Measure: Number; unit: percentage of participants
Groups:
- Safety: Safety population (treated patients)
Arm/Group | Safety
Number analyzed (Participants) | 5
percentage of participants
  TEAE Diarrhea | 80
  Serious Diarrhea | 0

ADVERSE EVENTS:
Time Frame: From time of first dose, through 28 days after last dose, assessed up to 16 months.
Description: Safety population: Participants receiving at least 1 dose of investigational product.
  Serious and Other Adverse Events were monitored/assessed only in the safety population
Arm/Group | Safety
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety (N=5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Faeces hard (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Paronychia (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT04366713/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04366713/SAP_001.pdf
  • Informed Consent Form (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04366713/ICF_002.pdf